CLINICAL TRIAL: NCT04506814
Title: Comparison of Repeat Endocardial PVI Vs Epicardial Posterior Wall Isolation and LAA Clip Plus PVI for Recurrent Atrial Fibrillation After Prior PVI
Brief Title: Endocardial Vs Epicardial Ablation for Recurrent Paroxysmal AF
Acronym: REPEAL-AF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding issues
Sponsor: University of Rochester (Other)
Collaborators: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Principal Investigator, Jonathan Steinberg, Collaborator, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UR Re-ablation Paroxysmal AF
Record Dates: First submitted 2020-08-04; First posted 2020-08-10 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Recurrent Paroxysmal Atrial Fibrillation Despite Prior Pulmonary Vein Isolation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Endocardial PVI (Active Comparator): Endocardial complete PVI
  Interventions: Device: Endocardial PVI
- Epicardial Posterior Wall Isolation + LAA Exclusion + Endocardial PVI (Experimental): Minimally invasive surgical hybrid ablation using the convergent approach plus LAA exclusion using the clip
  Interventions: Device: Epicardial Posterior Wall Isolation + LAA Exclusion + Endocardial PVI

INTERVENTIONS:
Device: Endocardial PVI — Catheter based PVI
  Arms: Endocardial PVI
Device: Epicardial Posterior Wall Isolation + LAA Exclusion + Endocardial PVI — Minimally invasive PVI with posterior wall RF ablation + LAA clip + endocardial PVI
  Arms: Epicardial Posterior Wall Isolation + LAA Exclusion + Endocardial PVI

SUMMARY:
There is no current accepted and predictably effective ablative therapy for patients with recurrent paroxysmal atrial fibrillation after prior pulmonary vein isolation (PVI). This study will compare redo PVI with hybrid epicardial ablation incorporating posterior wall isolation and LAA clip, and redo PVI.

DETAILED DESCRIPTION:
In these redo ablation patients, the ideal re-ablation strategy is unknown and many techniques have been proposed but there is no consensus nor strong clinical trial data.

This treatment gap prompted the development of a combined minimally invasive epicardial and endocardial ablation ("Convergent") procedure. During the last decade, this "hybrid" approach has garnered increasing acceptance in clinical practice, with several reports of promising antiarrhythmic outcomes in challenging disease states, as well as modifications to maximize safety and clinical outcomes. One key aspect of this approach is that it targets key drivers of AF including the PVs but also the left atrial posterior wall (LAPW), combining endocardial and epicardial energy delivery. The LAPW (or "PV myocardium") shares similar embryological origins and electrophysiological properties with the PVs, is predisposed to develop fibrosis, and thus recognized as an important source of AF. Recently, the CONVERGE randomized clinical trial demonstrated superiority of this hybrid approach compared to PVI in patients with persistent AF.

The left atrial appendage (LAA) has also been designated as a potential important trigger site of AF, and if isolated, may result in improved post-ablation AF outcomes. Although catheter-based isolation is controversial due to the potential to increase the risk of stroke, surgical exclusion of the LAA by placement of an occlusive clip has been suggested to be both antiarrhythmic and anti-thrombotic. Thus it is proposed in this trial to incorporate the LAA clip within the hybrid procedure.

Given the sheer volume of patients undergoing ablation of AF and the predictable necessity to perform repeat ablation procedures on a portion of these patients, the need for a proven redo ablation strategy is self-evident. The investigators thus propose a randomized clinical trial to determine if there is incremental efficacy by performing LAPW/LAA isolation via a hybrid approach in comparison to the conventional redo PVI alone in patients with paroxysmal AF.

ELIGIBILITY:
Inclusion Criteria

1. Age > 18 years
2. Symptomatic paroxysmal AF despite prior 1 or 2 PVI procedures within past 10 years (paroxysmal AF lasting up to 7 days before spontaneous termination)
3. Eligible for referral for re-ablation based on current guidelines
4. LA diameter < 6.0 cms on transthoracic echo
5. Willingness to comply with post-procedural follow-up requirements and to sign informed consent

Exclusion Criteria

1. Inability to undergo AF catheter ablation (e.g., presence of a left atrial thrombus, contraindication to anticoagulation)
2. Prior history of open heart surgery
3. Prior history of pericarditis or pericardiocentesis
4. Prior history of stroke/TIA/systemic embolism
5. NYHA class IV congestive heart failure or LVEF < 25%
6. Persistent or longstanding persistent AF (duration > 1 year)
7. Coronary revascularization or valve surgery within 3 months
8. Prior valve surgery using a mechanical prosthesis
9. An estimated glomerular filtration rate (eGFR) < 45mL/min/1.73m2, using the MDRD calculation
10. Life expectancy <1 year for any medical condition
11. AF due to reversible cause e.g. hyperthyroid state
12. Women who are pregnant or plan to become pregnant during the course of the trial** Note: Women of childbearing potential must have a negative pregnancy test within 7 days prior to randomization.
13. Participation in other clinical trials that will affect the objectives of this study
14. History of non-compliance to medical therapy
15. Inability or unwillingness to provide informed consent
16. Resides at such a distance from the enrolling site so travel to follow-up visits would be unusually difficult
17. Does not anticipate residing in the vicinity of the enrolling site for the duration of the trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation > 30 secs | At 1 year
  Based on serial 7-day Holter recordings

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Short Hills, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No